CLINICAL TRIAL: NCT01656031
Title: A Phase II Open-Label Study of High-Dose Cytarabine and Clofarabine in Adult Patients With Refractory or Relapsed Acute Myelogenous Leukemia or Refractory or Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21204 Phase 2; CCCWFU-21204; ILEX-CCCWFU-21204; CCCWFU-BG04-519
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-02

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- high-dose cytarabine and clofarabine (Experimental): high-dose cytarabine (2000 milligram/meter squared/day) administered intravenously over 3 hours followed by clofarabine administered intravenously over 2 hours daily for 5 consecutive days
  Interventions: Drug: clofarabine; Drug: cytarabine

INTERVENTIONS:
Drug: clofarabine
Drug: cytarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying clofarabine when given together with cytarabine to see how well they work in treating patients with refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in adult patients with relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia treated with high-dose cytarabine followed by clofarabine.

OUTLINE: This is an open-label phase II study. Patients are stratified according to diagnosis (acute myeloid leukemia vs acute lymphoblastic leukemia Phase II: Patients receive high-dose cytarabine followed by clofarabine (at the dose determined in phase I) on days 1-3.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 39 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologic confirmation of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL)

  * No M3 AML
* Meets 1 of the following criteria:

  * In first relapse
  * In second relapse after a second complete remission (CR) that lasted ≥ 3 months
  * Refractory to initial induction therapy
* No symptomatic CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 2
* Creatinine < 2 mg/dL
* Bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 4 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after completing study treatment
* Ejection fraction ≥ 45% by echocardiogram
* No active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant
* No psychiatric disorders that would interfere with giving consent, study participation, or follow-up procedures
* No other severe concurrent disease that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* At least 1 week since prior therapy and recovered
* No other concurrent chemotherapy

  * Hydroxyurea to control WBC count before starting study treatment allowed
* No concurrent corticosteroids unless used for diseases other than leukemia
* No concurrent palliative radiotherapy
* No concurrent growth factors (e.g., epoetin alfa, filgrastim [G-CSF], or sargramostim [GM-CSF]) in patients with AML

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayard L. Powell, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiment began 02/28/2005 and ended 08/06/2008.
Groups:
- High-dose Cytarabine and Clofarabine: high-dose cytarabine administered intravenously over 3 hours followed by clofarabine administered intravenously over 2 hours daily for 5 consecutive days
Period: Overall Study
Arm/Group | High-dose Cytarabine and Clofarabine
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High-dose Cytarabine and Clofarabine
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 27
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Measure Patient Response to High-dose Cytarabine Followed by Clofarabine in Adult Patients With Relapsed or Refractory AML
Description: Response to the therapy is measured by a defined improvement in Neutrophil and platlet counts, along with improved cellularity of bone marrow biopsy (>20% with maturation of all cell lines), <5% blasts, auer rods must not be detectable and extramedullary leukemia or soft tissue involvment must not be present.
Time Frame: 5 weeks
Measure: Number; unit: participants
Arm/Group | High-Dose Cytarabine and Clofarabine
Number analyzed (Participants) | 39
participants | 17

ADVERSE EVENTS:
Arm/Group | High-Dose Cytarabine and Clofarabine
Serious Adverse Events (participants affected / at risk) | 39/39
Other Adverse Events (participants affected / at risk) | 39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Cytarabine and Clofarabine (N=39)
low Platelets (Investigations) | 39 (39)
Low WBC (Investigations) | 39 (39)
Low ANC (Investigations) | 38 (38)
Low Hemoglobin (Investigations) | 37 (37)
hypokalemia (Investigations) | 26 (26)
Lymphopenia (Investigations) | 23 (23)
serum glutamic pyruvic transaminase (Investigations) | 23 (23)
serum glutamic oxaloacetic transaminase (Investigations) | 22 (22)
Infection with high grade neutropenia (Infections and infestations) | 15 (15)
hypophosphatemia (Investigations) | 14 (14)
hyperglycemia (Investigations) | 12 (12)
Acidosis (Investigations) | 11 (11)
Febrile neutropenia (Investigations) | 11 (11)
Hypoxia (Investigations) | 9 (9)
hyponatremia (Investigations) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
hyperbilirubinemia (Investigations) | 8 (8)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7)
hypocalcemia (Investigations) | 7 (7)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Lung Infection with high grade neutropenia (Infections and infestations) | 6 (6)
Bicarbonate serum-low (Investigations) | 6 (6)
Hypotension (Cardiac disorders) | 6 (6)
Pain: Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Lipase (Investigations) | 4 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 4 (4)
Alkalosis (Investigations) | 4 (4)
Partial Thromboplastin Time (Investigations) | 4 (4)
Infection - Other (Infections and infestations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Urinary Infection with high grade neutropenia (Infections and infestations) | 3 (3)
infection associated with Lymphopenia (Infections and infestations) | 3 (3)
hyperuricemia (Investigations) | 3 (3)
Confusion (General disorders) | 3 (3)
Edema: viscera (Vascular disorders) | 3 (3)
hyperkalemia (Investigations) | 3 (3)
hypoalbuminemia (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Blood Infection with high grade neutropenia (Infections and infestations) | 2 (2)
Urinary with low grade neutropenia (Infections and infestations) | 2 (2)
hemorrhage/bleeding into skin or mucosa (Skin and subcutaneous tissue disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 2 (2)
Colitis infectious (Infections and infestations) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
hypernatremia (Investigations) | 2 (2)
hypermagnesemia (Investigations) | 2 (2)
Fatigue (General disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 2 (2)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Anorexia (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
hypocalcemia (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Upper airway Infection with high grade neutropenia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Trachea Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Skin Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Nose Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Brain Infection with high grade neutropenia (Infections and infestations) | 1 (1)
Bone Infection with high grade neutropenia (Infections and infestations) | 1 (1)
"Hemorrhage, pulmonary/upper respiratory" (Vascular disorders) | 1 (1)
"Hemorrhage, Vagina" (Vascular disorders) | 1 (1)
"Hemorrhage, Bladder" (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
"Hemorrhage, Lung" (Vascular disorders) | 1 (1)
Pain: Rectum (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain: Esophagus (General disorders) | 1 (1)
functional obstruction of bowel (Gastrointestinal disorders) | 1 (1)
Hemorrhage Stomach (Blood and lymphatic system disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Face (General disorders) | 1 (1)
Death not associated with any term (General disorders) | 1 (1)
Pain: Chest wall (General disorders) | 1 (1)
Pain: Chest/thorax (General disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Iron overload (Investigations) | 1 (1)
Amylase (Investigations) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain: Abdomen (General disorders) | 1 (1)
Depression (General disorders) | 1 (1)
Mood alteration: Agitation (General disorders) | 1 (1)
Edema: limb (Vascular disorders) | 1 (1)
Edema: head and neck (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1)
hypomagnesemia (Investigations) | 1 (1)
hypoglycemia (Investigations) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | High-Dose Cytarabine and Clofarabine
Nausea (Gastrointestinal disorders) | 30/39 (30)
Vomiting (Gastrointestinal disorders) | 22/39 (22)
Diarrhea (Gastrointestinal disorders) | 31/39 (31)
Anorexia (General disorders) | 21/39 (21)
Alkaline phosphatase (Investigations) | 27/39 (27)
Creatinine (Investigations) | 17/39 (17)
Proteinuria (Investigations) | 8/39 (8)
Hair loss (General disorders) | 4/39 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13/39 (13)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 8/39 (8)
Hypertension (General disorders) | 6/39 (6)
Hypotension (Cardiac disorders) | 12/39 (12)
Neuropathy: sensory (Cardiac disorders) | 7/39 (7)
Pain (Nervous system disorders) | 4/39 (4)
Insomnia (General disorders) | 14/39 (14)
Rigors/chills (General disorders) | 15/39 (15)
Fatigue (General disorders) | 19/39 (19)
hyperglycemia (Investigations) | 27/39 (27)
hypoglycemia (Investigations) | 5/39 (5)
hypocalcemia (Investigations) | 27/39 (27)
hypomagnesemia (Investigations) | 30/39 (30)
hyponatremia (Investigations) | 18/39 (18)
hypokalemia (Investigations) | 12/39 (12)
Bicarbonate serum-low (Investigations) | 19/39 (19)
hypoalbuminemia (Investigations) | 31/39 (31)
hyperbilirubinemia (Investigations) | 19/39 (19)
serum glutamic pyruvic transaminase (Investigations) | 15/39 (15)
hypophosphatemia (Investigations) | 7/39 (7)
Constipation (Gastrointestinal disorders) | 8/39 (8)
Pain: Head/headache (General disorders) | 20/39 (20)
serum glutamic oxaloacetic transaminase (Investigations) | 16/39 (16)
hypermagnesemia (Investigations) | 5/39 (5)
hypernatremia (Investigations) | 18/39 (18)
Dysphagia (General disorders) | 4/39 (4)
Fever without neutropenia (General disorders) | 5/39 (5)
Urinary frequency/urgency (General disorders) | 6/39 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 9/39 (9)
Edema: limb (Vascular disorders) | 17/39 (17)
Edema: viscera (Vascular disorders) | 7/39 (7)
Confusion (Vascular disorders) | 8/39 (8)
Pruritus/itching (General disorders) | 6/39 (6)
Anxiety (General disorders) | 10/39 (10)
Depression (General disorders) | 7/39 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 18/39 (18)
Pain: Abdomen (Skin and subcutaneous tissue disorders) | 6/39 (6)
Partial Thromboplastin Time (Investigations) | 19/39 (19)
Pain: Joint (Investigations) | 5/39 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 13/39 (13)
Atrial fibrillation (Cardiac disorders) | 5/39 (5)
Pain: Back (General disorders) | 5/39 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4/39 (4)
Hemorrhage respiratory (Vascular disorders) | 4/39 (4)
Flatulence (Gastrointestinal disorders) | 4/39 (4)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7/39 (7)
Pain: Muscle (General disorders) | 4/39 (4)
Pain: Extremity-limb (General disorders) | 8/39 (8)
Pain: Skin (Skin and subcutaneous tissue disorders) | 5/39 (5)
Pericardial effusion (non-malignant) (Skin and subcutaneous tissue disorders) | 9/39 (9)
hemorrhage/bleeding into skin or mucosa (Cardiac disorders) | 5/39 (5)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 5/39 (5)
Sinus tachycardia (Cardiac disorders) | 14/39 (14)
Vitreous hemorrhage (Cardiac disorders) | 4/39 (4)
Psychosis (General disorders) | 5/39 (5)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 6/39 (6)
Conjunctiva with neutropenia (Eye disorders) | 3/39 (3)
Pain: Bone (General disorders) | 3/39 (3)
Ataxia (General disorders) | 3/39 (3)
hyperuricemia (Investigations) | 3/39 (3)
Dry mouth (General disorders) | 3/39 (3)
hyperkalemia (Investigations) | 3/39 (3)
hypercalcemia (Investigations) | 3/39 (3)
Taste alteration (General disorders) | 3/39 (3)
Dizziness (General disorders) | 3/39 (3)
Neuropathy: motor (Nervous system disorders) | 3/39 (3)
Stomatitis/Pharygitis (Infections and infestations) | 3/39 (3)
Hemorrhage/Bleeding - Other (Vascular disorders) | 3/39 (3)
Hemorrhage GU: Urinary (Vascular disorders) | 2/39 (2)
blurred vision (Eye disorders) | 2/39 (2)
Tremor (General disorders) | 2/39 (2)
Dental problems (General disorders) | 2/39 (2)
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 2/39 (2)
Supraventricular and nodal arrhythmia: Sinus arrhythmia (Cardiac disorders) | 2/39 (2)
photophobia (General disorders) | 2/39 (2)
Palpitations (Cardiac disorders) | 2/39 (2)
Osteonecrosis (Vascular disorders) | 2/39 (2)
Pain: Neck (General disorders) | 2/39 (2)
Muscle weakness (General disorders) | 2/39 (2)
Hemorrhage GI: Oral cavity (Vascular disorders) | 2/39 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 2/39 (2)
Pain: Chest wall (General disorders) | 2/39 (2)
Pain: Cardiac/heart (General disorders) | 2/39 (2)
Mood alteration: Agitation (General disorders) | 2/39 (2)
Heartburn/dyspepsia (General disorders) | 2/39 (2)
Edema: head and neck (Vascular disorders) | 2/39 (2)
Sweating (General disorders) | 2/39 (2)
Urinary retention (including neurogenic bladder) (General disorders) | 2/39 (2)
Low Hemoglobin (Investigations) | 2/39 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes